CLINICAL TRIAL: NCT07298694
Title: Improving Hypertension Management Through Preference List Defaults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Geisinger Clinic (Other)
Responsible Party: Principal Investigator, Gail Rosenbaum, Principal Investigator, Geisinger Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2025-0593
Record Dates: First submitted 2025-12-11; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Hypertension; Clinical Decision Support; Choice Behavior; Quality Improvement
Keywords: Hypertension; Clinical Decision Support; Choice Behavior; Quality Improvement
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Revised Preference List (Experimental): "(PREFERRED)" will be added to the beginning of the preference list for selected BP medications, which will frequently cause these medications to be listed first.
  Interventions: Behavioral: Revising preference list by adding "(PREFERRED)" to combination medication names
- No Change to the Preference List (No Intervention): Clinics will retain the usual EHR preference list order, with no changes to the default medication display.

INTERVENTIONS:
Behavioral: Revising preference list by adding "(PREFERRED)" to combination medication names — Providers in the intervention group will see "(PREFERRED)" listed before combination blood pressure medication names, which will frequently cause the combination medications to appear at the top of the EHR preference list.
  Arms: Revised Preference List

SUMMARY:
This study aims to evaluate whether modifying the EPIC preference list to display combination blood pressure (BP) medications at the top and/or adding "(PREFERRED)" to the beginning of the medication listing increases prescribing of these medications. Combination BP medications are aligned with value-based care guidelines and may improve patient adherence and reduce pill burden. Currently, these medications may be under-prescribed in part due to their low visibility in the EPIC prescribing interface.

DETAILED DESCRIPTION:
In this study, 50 primary care clinics at Geisinger will be randomized to a re-ordered preference list with combination BP medications at the top and/or adding "(PREFERRED)" to the beginning of the medication listing, or to have no change to the preference list.

This intervention works by adding a special character ( i.e., "(" ) to the beginning of a medication name in EPIC, which moves it to the top of the preference list. However, this only works when the provider searches for the first medication in a combination medication. For example, if a provider in the intervention group searches for "Amlodipine," the combination "(PREFERRED) Amlodipine-Benazepril" will appear at the top of the preference list.

However, a special character is NOT prioritized in the preference list when the second medication in a combination medication name is searched. For example, if the provider searches "Benazepril," the combination "(PREFERRED) Amlodipine-Benazepril" will be shown after single-class Benazepril prescriptions. The "(PREFERRED)" prefix will still be shown, which may encourage prescribing even without the medication listed first.

The study will employ a three-level hierarchical design, clustering patients within providers and providers within clinics. The study will run for 3 months or until enrollment reaches 12,150 unique patients, whichever comes second.

Clinic randomization will be stratified by variables that may affect response to the intervention including: clinic type (community medicine, senior medicine, internal medicine, FQHC), baseline prescribing rate for combination medications (<8%, 8%-13%, >13%), and number of providers (1-4, 5-9, 10-29, 30+).

One exception to the above stratification is internal medicine, where there are only two clinics. These are also the only two clinics with 30+ providers, but baseline combination medication prescribing rates fall in different stratification categories. These two clinics will be kept in the same stratum because they are still similar in culture, procedures, and size.

Stratified randomization was simulated 1000 times. Because strata are randomized independently and some strata include uneven numbers of clinics, overall assignment of the 50 clinics to treatment and control was uneven (e.g., 26 in treatment and 24 in control) on 709 of the 1000 iterations. To ensure a balance in clinic allocation to study arms, one of the 291 evenly randomized iterations will be randomly selected for implementation in the study.

ELIGIBILITY:
Inclusion Criteria:

* Order placed for a medication starting with any of the following: "amlodipine", "benazepril", "valsartan", "lisinopril", "hctz", "hydrochlorothiazide", "hydro", "losartan"
* The order is placed at an in-person, virtual (telemed), telephone, or nurse encounter in a clinic included in the study
* Patient is age 18+
* Order is placed in the clinician's primary clinic

Exclusion Criterion:

- Order was placed by a clinical leader who was aware of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12150 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Prescribing of Combination Antihypertensive Medication (y/n) | Day of the appointment (1 day)
  Defined as whether a provider prescribes a combination blood pressure medication (e.g., a single pill containing two medication classes) on the day of the patient's appointment. This is measured at the patient level using EHR prescribing data.

OTHER OUTCOMES:
Change in Systolic Blood Pressure | 6 months to 1 year after enrollment (whenever a qualifying reading is taken)
  Change in systolic blood pressure from baseline.
  If a reading was taken at the enrolling encounter, that reading will be used for baseline. If a reading was not taken at the enrolling encounter (e.g. because the encounter was virtual), the most recent qualifying reading in the 30 days prior to the encounter will be used.
  Follow-up readings for this outcome will be the first qualifying reading taken at least 6 months, but no more than 1 year, following the enrolling encounter.
  To qualify, readings taken outside the target encounter must be from non-acute outpatient encounters in primary care, nephrology, cardiology or endocrinology. If more than one reading was taken at the appointment, the last reading will be used.
  If the patient does not have a qualifying baseline and follow-up reading, they will be excluded from the analysis of this outcome.
Change in Diastolic Blood Pressure | 6 months to 1 year after enrollment (whenever a qualifying reading is taken)
  Change in diastolic blood pressure from baseline.
  If a reading was taken at the enrolling encounter, that reading will be used for baseline. If a reading was not taken at the enrolling encounter (e.g. because the encounter was virtual), the most recent qualifying reading in the 30 days prior to the encounter will be used.
  Follow-up readings for this outcome will be the first qualifying reading taken at least 6 months, but no more than 1 year, following the enrolling encounter.
  To qualify, readings taken outside the target encounter must be from non-acute outpatient encounters in primary care, nephrology, cardiology or endocrinology. If more than one reading was taken at the appointment, the last reading will be used.
  If the patient does not have a qualifying baseline and follow-up reading, they will be excluded from the analysis of this outcome.

IPD SHARING:
Plan to Share IPD: No